CLINICAL TRIAL: NCT01318044
Title: Thiopental Versus Propofol During Magnetic Resonance Imagining in Children
Brief Title: Thiopental Versus Propofol During Magnetic Resonance Imagining in Children: Something Old, Something New
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Antigona Hasani, University Clinical Center of Kosovo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCCK-30
Record Dates: First submitted 2011-03-11; First posted 2011-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-01

CONDITIONS: Complications
Keywords: thiopental; propofol; sedation; MRI
MeSH Terms: interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol group: propofol (Active Comparator)
  Interventions: Drug: Propofol and Thiopental
- Thiopental group: thiopental (Active Comparator)
  Interventions: Drug: Propofol and Thiopental

INTERVENTIONS:
Drug: Propofol and Thiopental — An initial bolus of 0.5 mg/kg of propofol will be administered over 1 minute. Supplementary boluses of propofol will be added until the UMSS score 3 are achieved.
  An initial bolus of 2 mg/kg of thiopental will be administered over 1 minute. Supplementary boluses of thiopental will be added until the UMSS score 3 are achieved
  Other Names: Diprivan; Nesdonal

SUMMARY:
Magnetic resonance imagining (MRI) in children requires sedation to achieve the degree of cooperation or immobilization, necessary to complete these procedures successfully. In this study the investigators analyze two most popular anesthetics used for this procedure, sodium thiopental and propofol. The aim of this study is to determine optimal dose of propofol and thiopental during MRI and to establish safety and efficacy of these drugs.

DETAILED DESCRIPTION:
This prospective, randomize, double-blind study will include 100 children, aged 6 month-12 years with ASA physical status I-II.

Children older than 3 years of age shall consume nothing by mouth (NPO) for solids and milk for at least 8 hours and children 6 months-3 years of age are NPO for solids and milk for 6 hours. Children will be allowed to receive breast milk until 4 hours before the beginning of the sedation. All the children will be allowed to take clear liquids up until 2 hours before the beginning of the sedation. To facilitate IV drug administration, EMLA cream will be applied on the dorsum of both hands 1 h before transfer to the preparation room.

Presedation behavior will be assessed on a 4-point scale, (by an anesthesiologist 1; who does not know which drug is administered): 1 = calm, cooperative; 2 = anxious but reasonable; 3 = anxious and not reasonable; 4 = crying or resisting. Categories 1 and 2 will be called "nondistressed behavior," and categories 3 and 4 will be defined as "distressed behavior." Patients will receive: group I; propofol 0.5 mg/kg or group II; thiopental 2.0 mg/kg, for anesthetic induction. After initial dose of the drug the sedation level of the children will be measured by the anesthesiologist 2 using the University of Michigan Sedation Scale (UMSS). The UMSS assigns a score of 0-4 based on the clinical assessment of the level of sedation as follows: 0 = awake and alert; 1 = minimally sedated: tired/sleepy, appropriate response to verbal conversation and/or sound; 2 = moderately sedated: somnolent/sleeping, easily aroused with light tactile stimulation or a simple verbal command; 3 = deeply sedated: deep sleep, arousable only with significant physical stimulation, and 4 = unarousable. Scores 3 will be accepted as procedural sedation and 4 will be accepted as deep sedation.

If a UMSS score of 3 will not be achieved after initial dose of propofol and thiopental, supplementary boluses of drugs will be added.

Mean arterial blood pressure (MAP), heart rate (HR), peripheral oxygen saturation (Spo2), and respiratory rate (RR) will be monitored continuously and be recorded at 5-min intervals during the study period by anesthesiologist 1. Patients will be allowed to breathe spontaneously without an artificial airway throughout the procedure. Oxygen will be administered via facemask.

Quality of the MRI will be evaluated by a radiologist using a three-point scale (1 = no motion; 2 = minor movement; 3 = major movement necessitating another scan).

Recovery time will be accepted as the period of time between the ends of MRI scan and reaching a UMSS score of 2 (by an anesthesiologist 2).

Side effects (apnea, nausea, vomiting, laryngospasm, emergence agitation) could occur during and after sedation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 6 months - 12 years old
* Patient is scheduled for MRI at University Clinical center of Kosovo
* Patients is ASA I/II
* Patient meets criteria to receive either propofol or thiopental sedation
* Patient's parent/guardian provides written consent

Exclusion Criteria:

* Patients with ASA > II
* Patients with airway abnormalities
* Patients with known allergies to the study drugs
* Parent/guardian refusal of participation

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
presedation behavior | day of sedation (day 1)
  Presedation behavior will be assessed on a 4-point scale, (by an anesthesiologist 1; who does not know which drug is administered): 1 = calm, cooperative; 2 = anxious but reasonable; 3 = anxious and not reasonable; 4 = crying or resisting. Categories 1 and 2 will be called "nondistressed behavior," and categories 3 and 4 will be defined as "distressed behavior."

SECONDARY OUTCOMES:
to determine optimal dose of propofol and thiopental during MRI | day of sedation (day 1)
  The UMSS assigns a score of 0-4 based on the clinical assessment of the level of sedation as follows: 0 = awake and alert; 1 = minimally sedated: tired/sleepy, appropriate response to verbal conversation and/or sound; 2 = moderately sedated: somnolent/sleeping, easily aroused with light tactile stimulation or a simple verbal command; 3 = deeply sedated: deep sleep, arousable only with significant physical stimulation, and 4 = unarousable. Scores 3 will be accepted as procedural sedation and 4 will be accepted as deep sedation.
UMSS score | day of sedation (day 1)
Side effects of sedation | day of sedation (day 1)
  Side effects (apnea, nausea, vomiting, laryngospasm, emergence agitation) could occur during and after sedation will be recorded.
recovery times | day of sedation (day 1)
  Recovery time will be accepted as the period of time between the ends of MRI scan and reaching a UMSS score of 2 (by an anesthesiologist 2).

CONTACTS AND LOCATIONS:
Overall Officials: Antigona Hasani, MD,MSC, Study Chair — Anesthesiology and Reanimation
Locations (1):
- University Clinical Center of Kosovo, Tirana, Kosovo, Albania

REFERENCES:
- [Background] 1. Malvija S, Voepel -Lewis T, Eldevik OP, Rockwell DT, Wong JH, Tait AR. Sedation and general anaesthesia in children undergoing MRI and CT: adverse events and outcomes. Br J A naesth 2000; 84: 743-8. 2. Malviya S, Voepel-Lewis T, Tait AR, Merkel S, Tremper K, Naughton N. Depth of sedation in children undergoing computed tomography: validity and reliability of the University of Michigan Sedation Scale (UMSS). Br J Anaesth. 2002 ;88:241-5. 3. Koroglu A, Teksan H, Sagir O, Yucel A, Toprak HI, Ersoy OM. A comparison of the sedative, hemodynamic, and respiratory effects of dexmedetomidine and propofol in children undergoing magnetic resonance imaging. Anesth Analg. 2006;103:63-7.